CLINICAL TRIAL: NCT07304323
Title: Transforming Rehabilitation: Personalised Care for a Better Quality of Life (PREPARE, Phase 2)
Brief Title: Prepare II - Predictive Model Training and External Validation
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Prepare II; Project 101080288 - PREPARE (Other Grant/Funding Number: EUROPEAN HEALTH AND DIGITAL EXECUTIVE AGENCY (HADEA))
Record Dates: First submitted 2025-11-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HIP AND KNEE OSTEOARTHRITIS
Keywords: total joint arthroplasty; osteoarthritis; total joint replacement; inpatient rehabilitation; predictive model; rehabilitation outcomes
MeSH Terms: conditions — Osteoarthritis | interventions — Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent total hip and/or knee arthroplasty for primary or secondary osteoarthirtis: Patients discharged directly to inpatient rehabilitation unit in the same hospital.
  Interventions: Other: Functional rehabilitation

INTERVENTIONS:
Other: Functional rehabilitation — Functional rehabilitation is standardized educational and physical therapy to restore physical and activities of daily living function before discharge.
  Pain management, blood management and iron diet are also provided based on standard conditions (e.g. patient-reported pain, postoperative day and hemoglobin levels).
  Other Names: Pain management; Blood management; Iron diet

SUMMARY:
The general aim of the project is training and testing a predictive model of inpatient rehabilitation stay after hip and knee replacement for osteoarthritis. This specific part focuses on data collection and analysis for the model validation.

DETAILED DESCRIPTION:
The following variables will be investigated to evaluate their predictive value towards length of rehabilitation stay (primary outcome), place of discharge, burden of care at discharge and/or functional recovery (secondary outcomes):

* Patient age at admission
* Patient sex
* Patient profession
* Living status (e.g. home or residential unit)
* Diagnosis
* Surgical procedure
* American Society of Anesthesiologists Score
* Body Mass Index before surgery
* Day of surgery
* Duration of surgery (minutes)
* Surgical access technique
* Surgical ward stay
* Pre-existing comorbidities
* Pharmacological treatment of pre-existing conditions
* Hemoglobin levels at inpatient rehabilitation admission
* Pain (Numeric Rating Scale) at inpatient rehabilitation admission
* Function - cognitive domains at inpatient rehab admission
* Barthel Index of Activities of Daily Living (ADL) at inpatient rehab admission
* Physiotherapic functional evaluations
* Rehabilitation program
* Function - cognitive domains at inpatient rehab discharge
* Inpatient rehabilitation stay
* Place of discharge
* Use of walking aids at discharge
* Need of assistance with the ADL at discharge
* Barthel Index of Activities of Daily Living at inpatient rehab admission

Due to retrospective study design, patients will not be recruited ex-novo and will be used data already stored in the internal databases.

Data retrieved from clinical records and other sets internal to the hospital will be collected on a dedicated Excel sheet and divided per section of interest (baseline, intervention, outcomes).

Data from 1710 patients who underwent total hip or knee replacement and subsequent inpatient rehabilitation in our hospital were collected, in the previous part of this project, to train the model.

In this second part, the same variables from 400 patients will be collected to test the model predictivity. Put together, these samples represent around 80% and 20% of the total population (2100) respectively, which is a common cohort distribution to test for validity.

To verify the validity (discrimination and calibration) of the newly developed prediction and stratification models, we will conduct a temporal external validation based on a sample of newly collected patients undergoing hip and knee at the same hospital but at a different point in time (2018, as compared to 2019 for the development sample).

To this aim, we plan to include a convenience sample of at least 400 patients: the sample size was determined based on a minimum sample size calculation, using Hoeffding's inequality (DOI: 10.1016/j.jspi.2012.09.013), which is sufficient to identify differences in performance smaller than 10% performance points with confidence higher than 95% (minimum sample size=390).

Basic modelling methodologies such as linear and logic regression will also be taken into consideration.

The best performing model for each outcome of interest will be finally selected.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for THR and TKR at IRCCS Galeazzi Orthopedic Institute in 2018 (any month) and subsequently discharged to inpatient rehabilitation in the same structure.
* Aged ≥18 years.
* International Classification of Disease, Ninth Revision, Clinical Modification (ICD-9CM) Diagnoses: 715.15, 16, 25, 26 (primary and secondary osteoarthritis of the hip and knee).
* ICD-9CM Surgical procedures: 81.51, 81.54 (total joint replacement of the hip and knee).

Exclusion Criteria:

* Age < 18 years (if any).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to inpatient rehabilitation unit after discharged from surgical ward.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Length of inpatient rehabilitation stay (days) | Up to 30 days
  The number of days needed by the patient to be discharged in safety

SECONDARY OUTCOMES:
Need of care at discharge | Last day of inpatient rehabilitation stay: up to 30 days
  Hours of care (number) needed by the patient (estimation) to receive support on the Activities of Daily Living after hospital discharge.
Place of discharge | Last day of inpatient rehabilitation stay: up to 30 days.
  Home, home with care givers, other inpatient unit.
Barthel Index of autonomy in Activities of Daily Living (ADL) | Last day of inpatient rehabilitation stay: up to 30 days.
  Score 0-100 in both scales.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Pennestrì, PhD, Principal Investigator — IRCCS Ospedale Galeazzi Sant'Ambrogio
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Researchers of the same facility will scan paper records to retrieve patient data.
  No sensitive data will leave the hospital.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol is already completed and available. Informed consent is given based on retrospective study policy guidelines from the Ministry of Health.
Access Criteria: The researchers employed on the project will have access to paper-scan clinical records in a pdf format, either from the internal, protected database, or from a Compact Disc record.
URL: https://www.grupposandonato.it/strutture/ospedale-galeazzi-sant-ambrogio/informativa-privacy-studi-retrospettivi